CLINICAL TRIAL: NCT05186558
Title: A Multi-center, Single-arm, Open Label Study to Assess the Efficacy and Safety of Anti-PD-1 Antibody (Penpulimab) Plus Lenalidomide, Rituximab, Gemcitabine and Oxaliplatin (R2-GemOx) in Patients With Relapsed/ Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: Penpulimab Plus R2-GemOx Regimen in Relapsed or Refractory DLBCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-SR-545
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Neoplasms by Histologic Type
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Neoplasms by Histologic Type | interventions — penpulimab; Lenalidomide; Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- penpulimab, lenalidomide, rituximab, gemcitabine and oxaliplatin（Penpulimab-R2-GemOx)） (Experimental): penpulimab: 200 mg q2w, iv, drip R2-GemOx: lenalidomide 10 mg，po; Rituximab 375mg/m2, iv, drip; Gemcitabine 1000mg, po; Oxaliplatin 100mg/m2, iv, drip;
  Interventions: Drug: penpulimab, lenalidomide, Rituximab, Gemcitabine, Oxaliplatin

INTERVENTIONS:
Drug: penpulimab, lenalidomide, Rituximab, Gemcitabine, Oxaliplatin — Patients receive penpulimab+R2-GemOx two weeks for a cycle, detailed as follows:
  Combination therapy Anti-PD-1 antibody (penpulimab): Fixed dose of 200 mg every 2 weeks, d0, intravenous drip (without pretreatment), for 6 cycles.
  R2-GemOx: lenalidomide 10 mg，d1-7; Rituximab 375mg/m2, d0; Gemcitabine 1000mg, d1; Oxaliplatin 100mg/m2, d1; every 2 weeks for a cycle, 6 cycles as protocol specified.
  Maintenance treatment:
  Combination of two drugs:
  * Anti-PD-1 antibody (penpulimab): Fixed dose of 200 mg every 2 weeks, d0, intravenous drip (without pretreatment), , for 6 months
  * lenalidomide: 10 mg, po, for 18 months.
  Other Names: lenalidomide; Rituximab; Gemcitabine; Oxaliplatin

SUMMARY:
This study evaluates the efficacy and safety of penpulimab plus lenalidomide, rituximab, gemcitabine and oxaliplatin (R2-GemOx) in patients with relapsed/refractory diffuse large B cell lymphoma (DLBCL). All patients will receive six cycles of penpulimab plus R2-GemOx. Afterwards, 1) patients who achieve complete response (CR)/unconfirmed (CRu)/partial response (PR) assessed by positron emission tomography/computedtomography (PET-CT) and are eligible for autologous stem cell transplantation (ASCT) will undergo ASCT. 2) Patients who achieve CR/CRu/PR assessed by PET-CT and are not eligible for ASCT will directly receive penpulimab and lenalidomide as maintenance treatment, penpulimab for a maximum of 6 months, lenalidomide monotherapy for 18 months. 3) Patients achieved stable disease (SD) or progression disease (PD) assessed by PET-CT will withdraw from this study and receive proper treatment based on investigator's decision.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed CD20+ diffuse large B-cell lymphoma
* Age range from 18 to 80 years;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
* Expectation survival time over 3 months;
* According to Lugano 2014, at least one measurable nodular lesion with a length of greater than 15 mm, or extranodal lesion greater than 10 mm, lesion on FDG-PET scan demonstrates uptake);
* Diffuse large B-cell lymphoma patients failed to first-line rituximab based chemotherapy including anthracycline or anthracycline
* Patients are allowed to receive palliative radiotherapy, but the last time radiotherapy cannot be within 7 days before the first study drug administration;
* Adequate organ function
* Willingness to provide written informed consent.

Exclusion Criteria:

* Pregnant or lactating women;
* Subjects with a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) in the past 12 months;
* Patients with autoimmune diseases requiring treatment or with a history of syndrome requiring systemic use of steroid immunosuppressive agents, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc;
* Patients received systemic glucocorticoid therapy (excluding nasal spray, inhaled or other topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days prior to the first administration;
* Uncontrolled heart disease, including unstable angina pectoris, acute myocardial infarction 6 months before randomization, congestive heart failure (NYHA) heart function grade III or IV; or left ventricular ejection fraction of the heart <50% ；
* Patients are allergic to penpulimab, lenalidomide, CD20 monoclonal antibody and GemOx regimen
* Patients who have had previous organ transplants (except autologous hematopoietic stem cell transplants);
* History of other malignancy within the past 5 years (except for 1. basal cell carcinoma of the skin and 2. carcinoma in situ of the cervix and 3. patients who had received treatment for the purpose of cure and had not developed a malignant tumor with a known active disease in the previous 5 years);
* Those who have had neurotoxicity of grade 3 or above within two weeks before treatment;
* Severe or uncontrolled infections;
* Patients with drug abuse, medical, psychological or social conditions that may interfere with the study results or the assessment of the study results;
* Patients are unsuitable for the enrollment according to investigator's judgement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 6 weeks after the last dose of the combination therapy (each cycle is 14 days)
  Complete response rate after treated by penpulimab and R2-GemOx

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  from date of inclusion to date of death from any cause
Progression-free survival（PFS） | 2 years
  from date of inclusion to date of progression, relapse, or death from any cause
Rate of grade 3 or 4 treatment related adverse effect | Up to 30 days after the last cycle of per-protocol treatment and 90 days after last dose of anti-PD-1 antibody
  All the adverse events of the patients related will be assessed and graded by NCI CTCAE v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)
Locations (4):
- China (4):
  - The First affiliated Hospital of AnHui Medical Universtiy, Hefei, Anhui
  - ChangZhou First People's Hospital, Changzhou, Jiangsu
  - Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu
  - The First Affiliated Hospital Of Nantong University, Nantong, Jiangsu

REFERENCES:
- [Derived] Liang JH, Xing TY, Gu WY, Yin H, Zeng QS, Du KX, Sibusiso L, Wu JZ, Li Y, Wang F, Gao R, Li JY, Shen HR, Wang L, Xu W. Penpulimab in combination with lenalidomide and R-GemOx regimen (R2-GemOx-PD1i) in relapsed or refractory diffuse large B-cell lymphoma: a multicenter, single-arm, phase 2 trial. BMC Med. 2026 Feb 9. doi: 10.1186/s12916-026-04679-1. Online ahead of print. PMID 41656201